CLINICAL TRIAL: NCT00003026
Title: Long Term Adjuvant Hormonal Treatment With LHRH Analogue Versus No Further Treatment in Locally Advanced Prostatic Carcinoma Treated by External Irradiation and a Six Months Combined Androgen Blockade - A Phase III Study
Brief Title: Hormone Therapy in Treating Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22961; EORTC-22961; EORTC-GU-22961
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Flutamide; Triptorelin Pamoate; Radiotherapy

INTERVENTIONS:
Drug: bicalutamide
Drug: flutamide
Drug: triptorelin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using triptorelin may fight prostate cancer by reducing the production of androgens.

PURPOSE: Randomized phase III trial to compare the effectiveness of long-term hormone therapy and triptorelin with no further treatment in treating patients who have advanced prostate cancer previously treated with radiation therapy and 6 months of androgen suppression.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the best hormonal scheme to be associated with pelvic radiotherapy in the curative management of prostatic carcinoma for hormonal treatment with regards to treatment outcome (overall survival, clinical disease free survival, local regional control), quality of life (treatment side effects, sexual function), and health economy (cost effectiveness ratio).

OUTLINE: This is a randomized, multicenter study.

Patients receive external radiation for 5 weeks, followed by a pelvic boost given for 2 weeks and a 6 month combined androgen blockage initiated at the onset of external irradiation. Flutamide (Eulexin) or bicalutamide (Casodex) may be used as the antiandrogens. Antiandrogen treatment starts 1 week before the first injection of triptorelin.

Patients are then randomized to one of two treatment arms.

* Arm I: Patients receive no further treatment.
* Arm II: Patients receive antiandrogen for 2.5 years plus and LHRH analogue (triptorelin) administered every 3 months. Patients then continue the LHRH analogue alone for an additional 2.5 years in the absence of disease progression.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 966 patients will be accrued over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * T1c-T2a-b, N1-2 or pN1-2 (after pelvic lymphadenectomy)
  * T2c-T4, N0-2
* Prior external radiotherapy for locally advanced prostatic carcinoma required
* Prior hormone therapy (6 months of combined androgen blockade) for locally advanced prostatic carcinoma required with PSA no greater than 150 ng/mL before administration
* No progressive disease after the 6 months of combined androgen blockage
* No stages T1c/T2a-b with a negative pelvic lymph nodes status that is assessed clinically or surgically
* No lymph node involvement to common iliac and/or periaortic lymph nodes (M1a)
* No external iliac lymph node metastasis more than 5 cm in greatest dimension (N3)
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* WHO 0-2

Life expectancy:

* At least 5 years

Hematopoietic:

* Hemoglobin at least 10 g/dL
* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior or concurrent cancers other than basal cell skin cancer
* No serious nonmalignant disease resulting in a life expectancy of less than 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for prostate cancer

Chemotherapy

* No prior chemotherapy for prostate cancer

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 966 (Estimated)
Dates: Start 1997-04; Primary Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bolla, MD, Study Chair — CHU de Grenoble - Hopital de la Tronche; T. M. de Reijke, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (17):
- Belgium (6):
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Hospital, Hasselt
  - U.Z. Gasthuisberg, Leuven
- Rambam Medical Center, Haifa, Israel
- St. Luke's Hospital and Medical School, Guardamangia, Malta
- Netherlands (6):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Elisabeth Ziekenhuis, Tilburg
- Medical Radiological Research Center, Obninsk, Russia
- Marmara University Hospital, Istanbul, Turkey (Türkiye)
- City General Hospital, Stoke-on-Trent, England, United Kingdom

REFERENCES:
- [Result] Bolla M, de Reijke TM, Van Tienhoven G, Van den Bergh AC, Oddens J, Poortmans PM, Gez E, Kil P, Akdas A, Soete G, Kariakine O, van der Steen-Banasik EM, Musat E, Pierart M, Mauer ME, Collette L; EORTC Radiation Oncology Group and Genito-Urinary Tract Cancer Group. Duration of androgen suppression in the treatment of prostate cancer. N Engl J Med. 2009 Jun 11;360(24):2516-27. doi: 10.1056/NEJMoa0810095. PMID 19516032
- [Result] Bolla M, van Tienhoven G, de Reijke TM, et al.: Concomitant and adjuvant androgen deprivation (ADT) with external beam irradiation (RT) for locally advanced prostate cancer: 6 months versus 3 years ADT--results of the randomized EORTC phase III trial 22961. [Abstract] J Clin Oncol 25 (Suppl 18): A-5014, 238s, 2007.
- [Result] Giraud JY, Dusserre A, Conil M, et al.: Results of the dummy-run of EORTC trial no.22961: a phase III study of long term hormonal treatment on locally advanced prostatic carcinoma treated by radiation therapy and a 6 months CAB. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-699, 378, 2001.
- [Derived] King MT, Chen MH, Collette L, Neven A, Bolla M, D'Amico AV. Association of Increased Prostate-Specific Antigen Levels After Treatment and Mortality in Men With Locally Advanced vs Localized Prostate Cancer: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2021 May 3;4(5):e2111092. doi: 10.1001/jamanetworkopen.2021.11092. PMID 33999161